CLINICAL TRIAL: NCT00002297
Title: A Multi-Center Double-Blind Placebo-Controlled Study to Investigate the Action of Isoprinosine (Inosiplex) in Patients With Unexplained Generalized Lymphadenopathy
Brief Title: A Study of Isoprinosine in Patients With Lymph Node Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newport Pharmaceuticals International (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 008A; ISO-103-USA
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-06

CONDITIONS: Lymphatic Disease; HIV Infections
Keywords: Inosine Pranobex; AIDS-Related Complex
MeSH Terms: conditions — Lymphatic Diseases; HIV Infections; AIDS-Related Complex | interventions — Inosine Pranobex

INTERVENTIONS:
Drug: Inosine pranobex

SUMMARY:
The objectives of this study are to determine the effects of isoprinosine in patients diagnosed as having unexplained generalized lymphadenopathy. Variables to be examined will include:

Signs and symptoms:

* Lymphadenopathy.
* Fever.
* Weight loss.
* Occurrence of opportunistic infections.

Cell-mediated immune system parameters:

* T-helper cell (OKT4) numbers and proportions.
* T-suppressor cell (OKT8) numbers and proportions.
* Natural killer (NK) cell activity.
* Lymphocyte blastogenic response to phytohemagglutinin (PHA).
* Lymphocyte blastogenic response to pokeweed mitogen (PWM).
* Immunoglobulin (IgG, IgA, IgM, IgE, IgD) profile.
* Circulating immune complexes. Infections characteristically associated with AIDS, such as Candida albicans, Pneumocystis carinii pneumonia, Cytomegalovirus, Herpes simplex, Cryptococcus, Histoplasma, Toxoplasma, Cryptosporidium, Mycobacterium avium- intracellulare, Legionella, and Isospora.

Safety parameters:

* Blood chemistry including serum uric acid (PurposeA-12).
* Complete blood count (CBC).
* Platelet count.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with a history of gout, uric acid urolithiasis, uric acid nephrolithiasis, renal dysfunction, or gastric ulceration are excluded.

Concurrent Medication:

Excluded:

* Systemic corticosteroids.
* Cytotoxic immunosuppressive agents.
* Radiotherapy.

Critically ill patients or those with CDC-defined AIDS are excluded.

Prior Medication:

Excluded within 1 month of study entry:

* Immunotherapy.

Patients with persistent generalized lymphadenopathy (PGL).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Newport Pharmaceuticals International Inc, Laguna Hills, California, United States